CLINICAL TRIAL: NCT05424679
Title: Piloting +Connection is Medicine / The Healing Spirits Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00020570; OT2HD107543 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Issue; Depressive Symptoms; Anxiety
Keywords: American Indians and Alaska Natives; COVID-19; Safety Planning Intervention; Mental Health
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This pilot intervention trial will utilize a randomized controlled design with 1:1 allocation to either the intervention or control group. Both intervention and control groups will receive individualized coping plans, facilitated connections to care, and COVID-19 safety messages. The intervention group will receive caring messages sent on a standardized schedule in addition to what the control group receives.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals randomized to the intervention group will receive an evidence-based tool (coping plan + two additional check-in calls or visits), up to three COVID-19 safety messages, information on and facilitated referrals to community support services (e.g., tribal behavioral health), and up to seven culturally responsive caring messages (i.e. Caring Contacts) from the research team over a period of three months.
  Interventions: Behavioral: Safety Planning Intervention; Behavioral: Caring Contacts
- Control group (Active Comparator): Individuals randomized to the control group will receive an evidence-based tool (coping plan + two additional check-in calls or visits), up to three COVID-19 safety messages, and information on and facilitated referrals to community support services (e.g., tribal behavioral health) from the research team over a period of three months.
  Interventions: Behavioral: Safety Planning Intervention

INTERVENTIONS:
Behavioral: Safety Planning Intervention — The Safety Planning Intervention is a brief intervention that directly targets suicide risk with demonstrated efficacy and is a recommended best practice for suicide prevention. The intervention aims to provide participants with an individualized set of steps that can be used progressively to both reduce risk and maintain safety when under particular stress. It also includes a series of brief telephone calls to revise the safety plan and facilitate connections to care. The study team will adapt the intervention to target a larger range of mental health distress.
Behavioral: Caring Contacts — Caring contacts is a cost and time effective suicide prevention intervention. It traditionally utilizes letters and postcards that are sent to an individual to remind them that they are cared about and that they matter. Research suggests that this intervention significantly reduces the likelihood of dying by suicide and suicide attempt over a person's lifetime. This intervention has the potential to reach more individuals at risk in the community. In this study, the research team will allow participants to receive these messages by postcard/MMS and will adapt the intervention to align with cultural values.
  Arms: Intervention group

SUMMARY:
This study aims to assess what benefit, if any, an individualized coping plan and facilitating connections to care through referral coordination in conjunction with culturally tailored caring messages, (herein called the +Connection is Medicine intervention (Navajo Nation study name; +CiM)/The Healing Spirits Program (White Mountain Apache Tribe Study Name; HSP) have on the mental health of American Indian (AI) youth and caregivers who were previously identified as having high levels of anxiety and depression as part of their participation in a cohort study called Project SafeSchools (NIH Grant No.: OT2HD107543).

DETAILED DESCRIPTION:
The investigators will conduct a Pilot Randomized Controlled Trial (RCT) among caregivers and youth (11-16 years old) who score at elevated risk of anxiety or depression. Participants will be recruited from the sample of individuals who have scored "at risk" on a mental health screening assessment tool in an ongoing cohort study, Project SafeSchools (NIH Grant No.: OT2HD107543). All persons who screen "at risk" will be approached for this pilot study using the study's standardized recruitment script. Parent/Caregiver participants and youth participants may be enrolled separately. All potential study participants will be screened for eligibility after going through the consent/assent process. This is to confirm that potential participants are still presenting with elevated mental health scores at the start of enrollment. For parent/caregiver participants, the screening will utilize the same assessments as those used in the Project SafeSchools cohort study. All youth participants will complete a version of the brief screening tool as well. The screening tool plus a set of additional questions related to the interventions will be administered at 30 days post consent, and again at 90 days post consent to all participants. These additional assessments are needed to understand the immediate impact of the intervention approaches. Additional participant data from the Project SafeSchools study will be analyzed to better understand symptoms prior to the pilot study enrollment, and as a longer-term outcome assessment for the pilot study. If promising, the results of this study will inform a future fully powered study to test these interventions at scale. This pilot intervention will utilize a randomized controlled design, in which both the intervention and control groups receive individualized coping plans, facilitated connections to care, and COVID-19 safety messages. The intervention group also will receive regular caring messages.

ELIGIBILITY:
Inclusion Criteria:

- All participants must be parents/caregivers or index youth enrolled in a cohort study called Project SafeSchools.

Adult participants

* Have elevated levels of mental distress as reported in a Project SafeSchools assessment.
* Agreement to be re-contacted for future research as part of their Project SafeSchools consent.
* Meeting symptom eligibility criteria at a screening assessment/baseline visit indicating mental distress.

Youth participants:

* Are 11-16 years old
* Agreement from parent/caregiver to be re-contacted for future research from their Project SafeSchools consent form.
* Meeting symptom eligibility criteria based on a self-report screening assessment/baseline visit indicating mental distress.

For the inclusion criteria, mental distress is defined as meeting eligibility cutoff scores on the following instruments:

Adult Participants

* General Distress (Kessler)
* Anxiety (PROMIS)
* Depression (CESDR-10)
* Recent Suicide Ideation (either CESDR-10 or Ideation Questionnaire)

Youth Participants:

* Depression (CESDR-10)
* Emotional Problems (SDQ Emotional Problems Subscale)
* Anxiety (SCARED)
* Recent Ideation (Ideation question on CESDR-10 or ideation questionnaire)

Exclusion Criteria:

* Inability to cognitively complete interventions and assessments

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Haroz, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (4):
- United States (4):
  - Johns Hopkins Center for American Indian Health - Chinle Site, Chinle, Arizona
  - Johns Hopkins Center for American Indian Health - Tuba City Site, Tuba City, Arizona
  - Johns Hopkins Center for American Indian Health - Whiteriver Site, Whiteriver, Arizona
  - Johns Hopkins Center for American Indian Health - Shiprock Site, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: No
INSERT

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Individuals randomized to the intervention group will receive an evidence-based tool (coping plan + two additional check-in calls or visits), up to three COVID-19 safety messages, information on and facilitated referrals to community support services (e.g., tribal behavioral health), and up to seven culturally responsive caring messages (i.e. Caring Contacts) from the research team over a period of three months.
  Safety Planning Intervention: The Safety Planning Intervention is a brief intervention that directly targets suicide risk with demonstrated efficacy and is a recommended best practice for suicide prevention. It is the same as the Control group.
  Caring Contacts: Caring contacts is a cost and time effective suicide prevention intervention. It traditionally utilizes letters and postcards that are sent to an individual to remind them that they are cared about and that they matter. Research suggests that this intervention significantly reduces the likelihood of dying by suicide and suicide attempt over a person's lifetime. This intervention has the potential to reach more individuals at risk in the community. In this study, the research team will allow participants to receive these messages by postcard/MMS and will adapt the intervention to align with cultural values.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 38 | 36
Youth Participants (Two of these youth are older than 18. Our study considered 'youth' to be any child of a parent from a different study, who was recruited into the current study, regardless of age. By this definition, two adult children are considered 'youth'. This distinction will be reflected in the sample sizes for the Baseline Characteristics, where we report age based on the pre-defined disaggregations, in Primary Outcome 2 (youth only), Secondary Outcome 2 (adult only), and Secondary Outcome 3 (youth only).) | 5 | 4
Adult Participants | 33 | 32
Completed | 21 | 27
Not Completed | 17 | 9

BASELINE CHARACTERISTICS:
Population: Two participants that fall between 18- 65 years old are adult children, as determined by recruitment eligibility. Those participants are considered 'youth' in results reporting. This distinction is reflected in the difference between sample sizes for age, reported by the pre-defined disaggregations, and Participant Flow, Primary Outcome 2 (youth only), Secondary Outcome 2 (adult only), and Secondary Outcome 3 (youth only), per study definitions of adult and youth.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (12.4) | 35.6 (10.1) | 35.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native American or American Indian | 32 | 28 | 60
  Other Indigenous Ancenstry | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Multiple Races | 1 | 0 | 1
  No Race Reported | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 36 | 74
Distress [Mean (Standard Deviation); unit: units on a scale] — 0-24 score range where a score of 13+ is considered high risk
  units on a scale | 8.56 (3.84) | 8.69 (4.42) | 8.62 (4.10)

OUTCOME MEASURES:

1. Primary Outcome: Group Differences in Mean Scores for Caregiver and Youth General Distress Over Time as Assessed by the Kessler Psychological Distress Scale
Description: The Kessler Psychological Distress Scale is a six item self-report questionnaire that gathers information about a person's psychological distress. 0-24 score range where a score of 13+ is considered high risk.
Time Frame: Baseline (0 months); Midline (1 month post-baseline); End-line (3 months post-Baseline)
Population: Includes youth and adult participants.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 38 | 36
score on scale
  Baseline | 8.56 (3.84) | 8.69 (4.42)
  Midline | 6.52 (4.55) | 8.0 (4.67)
  End-line | 6.33 (5.88) | 7.19 (4.38)

2. Primary Outcome: Group Differences in Mean Scores for Youth Emotional Problems Over Time as Assessed by the Strengths and Difficulties Questionnaire
Description: The SDQ is a self-report questionnaire that can be used with youth ages 11-17. The emotional symptoms subscale is used in the questionnaire, which consists of 5 items. The questionnaire uses a 0-10 score range where a score of 5+ is considered high risk.
Time Frame: Baseline (0 months); Midline (1 month post-baseline); End-line (3 months post-Baseline)
Population: Youth only. Two adult children are included in analysis (i.e., older than 18), which reflects the Participant Flow numbers but differs from the Baseline Characteristics numbers. One adult child is in each group.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Intervention Group: Individuals randomized to the intervention group will receive an evidence-based tool (coping plan + two additional check-in calls or visits), up to three COVID-19 safety messages, information on and facilitated referrals to community support services (e.g., tribal behavioral health), and up to seven culturally responsive caring messages (i.e. Caring Contacts) from the research team over a period of three months.
  Safety Planning Intervention: The Safety Planning Intervention is a brief intervention that directly targets suicide risk with demonstrated efficacy and is a recommended best practice for suicide prevention. It includes a series of brief telephone calls to revise the safety plan and facilitate connections to care. The study team will adapt the intervention to target a larger range of mental health distress.
  Caring Contacts: Caring contacts is a cost and time effective suicide prevention intervention. It traditionally utilizes letters and postcards that are sent to an individual to remind them that they are cared about and that they matter. Research suggests that this intervention significantly reduces the likelihood of dying by suicide and suicide attempt over a person's lifetime. This intervention has the potential to reach more individuals at risk in the community. In this study, the research team will allow participants to receive these messages by postcard/MMS and will adapt the intervention to align with cultural values.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 5 | 4
score on scale
  Baseline | 5.75 (0.96) | 5.0 (2.65)
  Midline | 1.67 (1.15) | 4.33 (2.52)
  End-line | 3.0 (1.41) | 4.5 (4.95)

3. Secondary Outcome: Group Differences in Mean Scores for Caregiver and Youth Depressive Symptoms Over Time as Assessed by the Center for Epidemiologic Studies Depression Scale-Revised-10
Description: The CESDR-10 is a revised 10 item self-report questionnaire which measures depressive symptoms in general populations. It utilizes a 0-30 score range, in which a score of 8+ is considered high risk. The CESDR-10 also has one item that asks about recent suicide ideation.
Time Frame: Baseline (0 months); Midline (1 month post-baseline); End-line (3 months post-Baseline)
Population: Adult + Youth
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 38 | 36
score on scale
  Baseline | 10.9 (4.97) | 12.8 (6.01)
  Midline | 7.36 (5.92) | 10.4 (5.66)
  End-line | 6.62 (4.75) | 9.74 (6.54)

4. Secondary Outcome: Group Differences in Mean Scores for Caregiver Anxiety Over Time as Assessed by the Patient-Reported Outcome Measurement Information System
Description: PROMIS is an eight-statement survey that measures emotional distress due to anxiety that has been experienced over the previous seven days. It uses a five-point Likert scale, 1 indicating 'never' to 5 indicating 'always'. The survey is scored from 8-40 with a score of 17+ indicating high risk.
Time Frame: Baseline (0 months); Midline (1 month post-baseline); End-line (3 months post-Baseline)
Population: Adult caregivers only. The number of participants analyzed here matches the Participant Flow but differs from the Baseline Characteristics. The Baseline Characteristics age disaggregations include two adult children who our study considers as 'youth'. Therefore, the number reported here excludes these adult children.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 33 | 32
score on scale
  Baseline | 20.5 (5.32) | 20.6 (4.94)
  Midline | 16.7 (7.92) | 18.3 (6.51)
  End-line | 14.9 (6.69) | 15.8 (6.19)

5. Secondary Outcome: Group Differences in Mean Scores for Youth Anxiety Over Time as Assessed by the Screen for Child Anxiety Related Emotional Disorders
Description: The SCARED survey can be used with those aged 8-18 years. It includes 41 items and five scales which measure somatic/panic, general anxiety, separation anxiety, social phobia, and school phobia. SCARED uses a 0-82 score range where a score of 25+ is high risk.
Time Frame: Baseline (0 months); Midline (1 month post-baseline); End-line (3 months post-Baseline)
Population: Youth only. The number of participants analyzed matches the Participant Flow but differs from the Baseline Characteristics. Our study considered 'youth' to be children of parents from another study, regardless of age. Therefore, there are two adult children included in the Baseline Characteristics that we consider 'youth' and are reporting as such. One adult child is included in each intervention arm reported here.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 5 | 4
score on scale
  Baseline | 23.8 (8.62) | 26.7 (8.33)
  Midline | 9.0 (5.0) | 23.3 (19.9)
  End-line | 12.5 (13.4) | 20.0 (5.66)

6. Other Pre Specified Outcome: Group Differences in Mean Scores for Caregiver Social Connectedness Over Time as Assessed by a Subset of Questions That Measure Connection to Others and Several From the Communal Mastery Scale
Description: Investigators developed 4 items that measure connection to peers and family for use in the study. The Communal Mastery scale measures problem solving through the participant's community and social network. Three items from the Communal Mastery scale relevant to the intervention are included. All seven items are scored on a four-point Likert-type scale, with total possible range from 7-28. Higher scores represent higher levels of connectedness.
Time Frame: Baseline-3-months post-baseline; secondary data analysis to measure trends over 12-18 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Group Differences in Mean Scores for Caregiver and Youth Coping Behaviors Over Time as Assessed by a Subset of Questions From the Brief COPE Inventory
Description: 8 items out of 28 items in the brief COPE that are relevant to the intervention, focusing on coping behaviors that could be modified through the coping plan. Items are answered on a Likert-type scale. For this study, scores can range from 8 to 32 with higher scores representing higher levels of coping behavior.
Time Frame: Baseline-3-months post-baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Group Differences in Mean Scores for Youth Resilience Over Time as Assessed by Two Items From the Child/Youth Resilience Scale
Description: Two items related to social connections from the Child/Youth Resilience Scale were selected to assess youth resilience. Each question is rated on a scale of 1-5, for an overall scale score of 2-10. Higher scores represent a better outcome of more youth resilience.
Time Frame: Baseline-3-months post-baseline; secondary data analysis to measure trends over 12-18 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Group Differences in Youth Self-harm Scored as Individual Indicator Variables on Two Internally Developed Items
Description: Two items related to self-harm that were internally developed by the study team. The first item is answered yes or no. The second item asks about recency if the first item is yes. These items will be treated as indicator variables and will not be scored as a scale.
Time Frame: Baseline-3-months post-baseline; secondary data analysis to measure trends over 12-18 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Group Differences in Means Scores for Youth Knowledge of Coping Strategies as Assessed by One Internally Developed Item
Description: One item related to knowledge of coping strategies was internally developed by the study team. Items are scored using a Likert-type scale, with 0 indicating strong disagreement with a statement and 5 indicating strong agreement with a statement. Higher scores on this item will indicate more knowledge of coping strategies.
Time Frame: Baseline-3-months post-baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Group Differences in Caregiver and Youth Mental Health Service Knowledge, Access, and Use Scored as Individual Indicator Variables on an Internally Developed Questionnaire
Description: This is an internally developed questionnaire that includes 1 item on knowledge of mental health services in the community, 1 item on accessibility of mental health resources, 1 item on use of services in the previous 30 days, and 1 item on difficulties accessing services in the previous 30 days. The items on knowledge of services and accessibility of services are scored using a Likert-type scale, with 0 indicating strong disagreement with the statement and 5 indicating strong agreement with the statement. Items will be scored separately, with higher scores on each item indicating greater knowledge or accessibility. The two items on services use in the previous 30 days and difficulties accessing services in the previous 30 days use a single dichotomous answer (yes or no). These items will be analyzed separately with a dichotomous variable with yes representing service use or difficulties with service use in the past 30 days.
Time Frame: Baseline-3-months post-baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Group Differences in Average Scores for Caregiver and Youth COVID-19 Behaviors and Attitudes as Assessed by an Internally Developed Questionnaire
Description: This is an internally developed, 7-item inventory on participants' attitudes towards specific COVID-19 related behaviors, including masking, testing, and vaccinations. Scale scores range from 0-28, with higher score representing more positive attitudes towards COVID-19 prevention behaviors and attitudes.
Time Frame: Baseline-3-months post-baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected between baseline and end-line, a 9-month period.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/38 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT05424679/Prot_SAP_000.pdf